CLINICAL TRIAL: NCT00001061
Title: A Phase II, Double-Masked, Randomized, Placebo-Controlled Evaluation of Standard Therapy vs. Standard Therapy Combined With Human Monoclonal Anti-Cytomegalovirus Antibody (MSL 109) in the Therapy of AIDS Patients With Cytomegalovirus (CMV) Retinitis
Brief Title: Comparison of Two Methods in the Treatment of Cytomegalovirus of the Eyes in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Facet Biotech (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 266; 11242 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Foscarnet; Acquired Immunodeficiency Syndrome; Antibodies, Monoclonal; Cytomegalovirus Retinitis
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — sevirumab; Foscarnet; Ganciclovir

INTERVENTIONS:
Drug: Sevirumab
Drug: Foscarnet sodium
Drug: Ganciclovir

SUMMARY:
To evaluate the effect of MSL 109, human monoclonal anti-cytomegalovirus (CMV) antibody, on time to progression of CMV retinitis. To determine the safety and pharmacokinetic profile of MS 109. To evaluate the relationship between pharmacokinetic measurements of MSL 109 and efficacy and virologic markers.

Therapeutic agents currently available for CMV retinitis are limited by their inherent toxicities and short half-lives which require frequent intravenous dosing. Alternatively, MSL 109 has demonstrated safety and effectiveness in neutralizing CMV isolates at concentrations easily maintained in AIDS patients.

DETAILED DESCRIPTION:
Therapeutic agents currently available for CMV retinitis are limited by their inherent toxicities and short half-lives which require frequent intravenous dosing. Alternatively, MSL 109 has demonstrated safety and effectiveness in neutralizing CMV isolates at concentrations easily maintained in AIDS patients.

Patients receive induction therapy with intravenous ganciclovir or foscarnet daily for 14 days, then are placed on standard maintenance therapy with the induction drug for at least 11 months or until progression. Patients are randomized to receive 1 of 2 doses of MLS 109 or placebo every 2 weeks during induction and maintenance. They are followed at weeks 2 and 4 and every 4 weeks thereafter for 40 weeks. Patients who have not progressed by week 40 continue study drug with follow-up every 2 months until CMV progression occurs. AS PER AMENDMENT 11/29/96: Enrollment onto the current study has been discontinued. To study the enhancement of humoral immunity, a high-dose cohort has been added. Patients are now randomized to MSL 109 given at a higher dose or placebo administered at the same intervals as before. Randomization is weighted 2:1 in favor of high-dose MSL 109. Interim analyses will be performed to provide for early discontinuation, as indicated. Patients randomized under earlier versions may continue on their original study assignment if a study endpoint has not been reached.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* G-CSF and GM-CSF.
* Antiretroviral therapy.

Patients must have:

* HIV infection.
* First episode of CMV retinitis.
* No prior end-organ CMV disease - PER AMENDMENT 4/25/96: No prior end organ CMV disease within the past 6 months. Subjects who have been prophylaxed with oral ganciclovir and develop an episode of CMV retinitis are eligible.
* No active AIDS-defining opportunistic infection or malignancy that requires nephrotoxic or myelosuppressive therapy.
* Life expectancy of at least 6 months.
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* This protocol is approved for prisoner participation.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* PER AMENDMENT 4/25/96: Retinal detachment not scheduled for surgical repair, in all eyes meeting other eligibility criteria. (Was written as - No current retinal detachment (although old retinal detachments unrelated to HIV infection which have been repaired are permitted).
* Corneal, lens, or vitreous opacification that precludes funduscopic exam.
* Clinically significant pulmonary or neurologic impairment, such as intubation or coma. (Patients with a CNS mass or history of seizure disorder may enroll.)
* Tuberculous, diabetic, or hypertensive retinopathy, or other retinal lesions that would interfere with measurements of response or progression.
* Known hypersensitivity to the study drugs.

PER AMENDMENT 4/25/96:

* Presence of CMV retinal lesions that are only in areas of the retina which cannot be photographed.

Concurrent Medication:

Excluded:

* Immunomodulators, biologic response modifiers, interferon, or investigational agents that may influence course of CMV infection.
* Systemic acyclovir or any nephrotoxic agent, specifically aminoglycosides, amphotericin B, and parenteral pentamidines.
* Any concomitant therapy that would preclude use of cidofovir, foscarnet or ganciclovir.

Prior Medication:

Excluded: PER AMENDMENT 4/25/96:

* Use of IV ganciclovir, foscarnet or cidofovir within 6 months prior to study enrollment. (Was written - Ganciclovir or foscarnet for non-CMV herpes infections within 6 months prior to study entry.)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167
Dates: Study Completion 1998-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pollard RB, Study Chair; Borucki M, Study Chair; Gnann J, Study Chair; Hirsch MS, Study Chair
Locations (20):
- United States (20):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - Stanford CRS, Stanford, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Borucki M, Spritzler J, Gnann J, Hirsch M, Nokta M, Aweeka F, Pollard R. A phase II double masked, placebo-controlled evaluation of standard therapy vs standard therapy combined with human monoclonal anti-cytomegalovirus antibody (MSL-109) in the therapy of AIDS patients with newly diagnosed cytomegalovirus (CMV) retinitis in ACTG 266. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:154 (abstract no 460)
- [Background] CMV retinitis study aborted. GMHC Treat Issues. 1996 Sep;10(9):8. PMID 11363844
- [Result] Borucki MJ, Spritzler J, Asmuth DM, Gnann J, Hirsch MS, Nokta M, Aweeka F, Nadler PI, Sattler F, Alston B, Nevin TT, Owens S, Waterman K, Hubbard L, Caliendo A, Pollard RB; AACTG 266 Team. A phase II, double-masked, randomized, placebo-controlled evaluation of a human monoclonal anti-Cytomegalovirus antibody (MSL-109) in combination with standard therapy versus standard therapy alone in the treatment of AIDS patients with Cytomegalovirus retinitis. Antiviral Res. 2004 Nov;64(2):103-11. doi: 10.1016/j.antiviral.2004.06.012. PMID 15498605